CLINICAL TRIAL: NCT07382011
Title: Assessment of Craniofacial and Postural Changes Induced by LM-Activator Therapy in Growing Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haner Direskeneli, Principal investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarmaraLM
Record Dates: First submitted 2025-12-06; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Myofunctional Therapy; Orthodontic Appliance; Malocclusion Class II
Keywords: Myofunctional therapy; LM-Activator™; Cervical posture; Twin block appliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-Activator™ Therapy Group (Experimental): Children aged 8-13 years with Class II malocclusion received LM-Activator™ treatment. Skeletal, dentoalveolar, and cervical posture changes were evaluated prospectively.
  Interventions: Device: LM-Activator™
- Twin Block Appliance Group (Active Comparator): Children aged 8-13 years with Class II malocclusion treated with Twin Block appliances (archived records). Outcomes were analyzed for comparison with the experimental group.
  Interventions: Device: Twin Block Appliance

INTERVENTIONS:
Device: LM-Activator™ — The LM-Activator™ is a prefabricated myofunctional orthodontic appliance designed for early treatment of Class II malocclusion in growing children. In this study, children aged 8-13 years received LM-Activator™ therapy, and changes in skeletal, dentoalveolar, and cervical posture parameters were evaluated using cephalometric analysis and digital dental models.
  Arms: LM-Activator™ Therapy Group
Device: Twin Block Appliance — Twin Block is a removable functional appliance commonly used in the management of Class II malocclusion in children.
  Arms: Twin Block Appliance Group

SUMMARY:
This prospective study will compare the effects of LM-Activator™ and Twin Block appliances in 26 children (aged 8-13 years) with Class II malocclusion. Skeletal, dentoalveolar, and cervical posture parameters will be assessed using lateral cephalometric radiographs and digital dental models.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 8-13 years
* Cooperative behavior rated as "positive" or "definitely positive" according to the Frankl Behavior Rating Scale
* Presence of Class II malocclusion
* Patient-reported complaint of protruding anterior teeth
* Provision of written informed consent by both the child and their parent/legal guardian

Exclusion Criteria:

* Inability to continue treatment in the dental chair due to lack of cooperation
* Failure to attend scheduled follow-up appointments or withdrawal of consent during the study
* Occurrence of treatment-related complications preventing continuation of therapy (e.g., inability to maintain cooperation between patient and clinician)
* Inability to attend regular follow-up sessions or repeated absence from scheduled visits

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Overjet (mm) Assessed by Cephalometric Analysis | Up to 12 months
  Overjet defined as the horizontal distance (in millimeters) between the incisal edge of the maxillary and mandibular central incisors, measured on standardized lateral cephalometric radiographs. The outcome is calculated as the change from baseline to post-treatment.

SECONDARY OUTCOMES:
Change in ANB Angle (degrees) Assessed by Cephalometric Analysis | Up to 12 months
  ANB angle measured in degrees on standardized lateral cephalometric radiographs to evaluate the sagittal skeletal relationship between the maxilla and mandible. The outcome is calculated as the change from baseline to post-treatment.
Change in Overbite (mm) Assessed by Cephalometric Analysis | Up to 12 months
  Overbite defined as the vertical overlap (in millimeters) between the maxillary and mandibular central incisors, measured on standardized lateral cephalometric radiographs. Change calculated from baseline to post-treatment.
Change in SNA Angle (degrees) Assessed by Cephalometric Analysis | Up to 12 months
  SNA (Sella-Nasion-A point) angle measured in degrees on standardized lateral cephalometric radiographs to evaluate sagittal position of the maxilla relative to the cranial base. Change calculated from baseline to post-treatment.
Change in SNB Angle (degrees) Assessed by Cephalometric Analysis | Up to 12 months
  SNB (Sella-Nasion-B point) angle measured in degrees on standardized lateral cephalometric radiographs to evaluate sagittal position of the mandible relative to the cranial base. Change calculated from baseline to post-treatment.
Change in Upper Incisor Inclination (U1-SN, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  U1-SN angle measured in degrees on standardized lateral cephalometric radiographs to assess maxillary incisor inclination relative to the SN plane. Change calculated from baseline to post-treatment.
Change in Lower Incisor Inclination (IMPA, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  IMPA (Incisor Mandibular Plane Angle) measured in degrees on standardized lateral cephalometric radiographs to assess mandibular incisor inclination relative to the mandibular plane. Change calculated from baseline to post-treatment.
Change in Mandibular Plane Angle (Go-Me to SN, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  Mandibular plane angle measured in degrees as the angle between the Go-Me line and the SN plane on standardized lateral cephalometric radiographs (vertical skeletal pattern). Change calculated from baseline to post-treatment.
Change in Frankfort-Mandibular Plane Angle (FMA, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  FMA measured in degrees on standardized lateral cephalometric radiographs to assess vertical skeletal pattern. Change calculated from baseline to post-treatment.
Change in Jarabak Ratio (%) Assessed by Cephalometric Analysis | Up to 12 months
  Jarabak ratio calculated as a percentage from standardized lateral cephalometric radiographs to assess vertical facial proportions. Change calculated from baseline to post-treatment.
Change in Cranio-Cervical Angle (NSL-CVT, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  NSL-CVT angle measured in degrees on standardized lateral cephalometric radiographs to assess head and cervical posture (cranial base to cervical vertebra tangent). Change calculated from baseline to post-treatment.
Change in Cranio-Cervical Angle (NSL-OPT, degrees) Assessed by Cephalometric Analysis | Up to 12 months
  NSL-OPT angle measured in degrees on standardized lateral cephalometric radiographs to assess head posture relative to the odontoid process tangent. Change calculated from baseline to post-treatment.
Change in Inner Angle (degrees) Measured on Digital Dental Models | Up to 12 months
  Inner angle measured in degrees on digital dental models as defined in the study protocol. Change calculated from baseline to post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Recep Tayyip Erdoğan Külliyesi Sağlık Yerleşkesi, Diş Hekimliği Fakültesi, Başıbüyük Yolu 9/3 34854 Başıbüyük / Maltepe / İSTANBUL, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including intraoral photographs and clinical evaluation scores) may be shared in scientific publications or presentations. Data will be limited to information relevant for scientific analysis and will not include any personal identifiers.